CLINICAL TRIAL: NCT06967259
Title: A Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ENA-001 Administered as Intravenous (IV) and Intramuscular (IM) Doses
Brief Title: ENA-001 for Opioid Induced Respiratory Depression
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enalare Therapeutics Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENA-001-109; 4R44DA057133-02 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-05-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: The study protocol is an 8-period ascending, repeated, single dose, safety and tolerability study comparing the effects of ENA-001 with placebo in 4 panels of screened healthy volunteers after single doses. The study periods will be conducted for IV (4-periods) and for IM dosing (4-periods). The study will be randomized, double-blinded, and placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind for treatment but not dose level. The research pharmacist at the study center will not be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENA-001 Treatment Arm (Experimental): ENA-001 for intravenous injection will be given over 3-5 seconds and will be administered via a suitable arm vein with an indwelling catheter.
  ENA-001 for intramuscular injection will be administered over 3-5 seconds via both deltoid muscles.
  Interventions: Drug: ENA-001
- Placebo Treatment Arm (Placebo Comparator): Placebo for intravenous injection will be given over 3-5 seconds and will be administered via a suitable arm vein with an indwelling catheter.
  Placebo for intramuscular injection will be administered over 3-5 seconds via both deltoid muscles.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: ENA-001 — Concentration for ENA-001 IV formulation is 10 mg/mL. Concentration for ENA 001 IM formulation is 30 mg/mL.
  Arms: ENA-001 Treatment Arm
Drug: Placebo Comparator — Placebo comes in 5 mL/vial. Placebo matches ENA-001 injection; however, no ENA-001 is included.
  Arms: Placebo Treatment Arm

SUMMARY:
This study is a Phase I clinical trial to assess the safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) profiles with single intravenous (IV) and intramuscular (IM) doses of ENA-001.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing to give written informed consent for the trial and able to adhere to dose and visit schedules.
2. Male and female, >18 to ≤55 years of age.
3. Subject must weigh ≥50 to ≤100 kg.
4. Subjects must have Body Mass Index [weight/height2 (kg/m2)] between 18 to 30 kg/m2 (inclusive).
5. Have no clinical or electrocardiographic signs of ischemic heart disease as determined by the Investigator with normal cardiac intervals appropriate for their gender. The Screening 12 lead electrocardiogram (ECG) conduction intervals must be within gender specific normal range (e.g., QTcf female < 450 msec QT corrected for heart rate by Fridericia's cube root formula (QTcF) males < 430 msec, PR interval ≤ 220 msec). ECGs are to be judged by the investigator or sub-investigator as per standardized procedures.
6. Subjects' clinical laboratory tests (blood hematology, blood chemistry, coagulation and urinalysis and liver enzymes must be in normal range. Where applicable, normal range is defined as in the FDA guidance Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials.
7. Vital sign measurements must be within the following ranges during screening and on Day -1:

   1. body temperature, >35.5 C to ≤37.5 C
   2. systolic blood pressure, >90 to ≤140 mmHg
   3. diastolic blood pressure, >40 to ≤95 mmHg
   4. pulse rate, >55 to ≤100 bpm
8. Non-vasectomized men must agree to use a condom with spermicide (when marketed in the country), double-barrier contraception, abstain from heterosexual intercourse, or have a sole sexual partner of non-childbearing potential during the trial and for 3 months after stopping the medication. Male subjects must agree not to donate sperm from the time of dosing until 90 days after dosing.
9. Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have a negative pregnancy test prior to enrollment as well as prior to each subsequent period of dosing administration, and must agree to at least one of the following contraception requirements from screening through at least 3 months after the last dose of study drug:

   1. Be sexually inactive (abstinent)
   2. Hormonal or non-hormonal intrauterine device in place for at least 3 months prior to dosing with a barrier method (condom or diaphragm) and spermicide at least 3 months after last dose of study drug.
   3. Double barrier methods (e.g., condom and diaphragm) with spermicide for at least 30 days prior to screening and through at least 3 months after last dose of study drug. Hormonal oral contraception + use of condoms and spermicides is an acceptable double barrier method.
   4. Surgical sterilization of the partner (vasectomy at least six months prior to dosing) with a barrier method (e.g., condom or diaphragm) and spermicide through at least 3 months after last dose of study drug.
   5. Female subjects who claim to be sexually inactive but become sexually active during the course of the study must agree to use a double barrier method (e.g., condom and diaphragm) with spermicide from the time of the start of sexual activity through at least 3 months after last dose of study drug.

      In addition, female subjects of childbearing potential must be advised to remain sexually inactive or to keep the same birth control method through at least 3 months after last dose of study drug.

      Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to dosing:
      * Hysteroscopic sterilization and using a barrier method (e.g., condom or diaphragm) and spermicide throughout the study.
      * Bilateral tubal ligation or bilateral salpingectomy and be using a barrier method (e.g., condom or diaphragm) and spermicide throughout the study.
      * Hysterectomy.
      * Bilateral oophorectomy.
   6. Women with amenorrhea for at least 1 year prior to dosing and who have follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status, are considered post-menopausal and therefore of non childbearing potential.
10. Subjects must demonstrate a normal Allen's test for both hands, to assure adequate arterial collateral circulation.
11. Subjects must be free of any clinically significant disease that would interfere with the study evaluations.

Exclusion Criteria:

1. Current diagnosis of psychiatric disease requiring daily medication, including controlled or uncontrolled schizophrenia and current or recently treated depressive disorders.
2. Current diagnosis of Generalized Anxiety Disorder (DSM-5) requiring treatment.
3. History of alcohol abuse (more than an average of two (2) drinks per day) within the past two (2) years.
4. History of drug abuse within the past two years.
5. History of regular smoking/vaping or any use of nicotine products within the past year (>5 per week means exclusion).
6. Failure to take or test positive of the drug of abuse tests or alcohol urine test at screening or check-in.
7. Positive for HIV, or Hepatitis B or C at screening.
8. Blood donation or blood loss within 60 days of screening or plasma donation within 7 days of screening.
9. Subjects with a history of bleeding disorders or coagulopathies.
10. History of dyspnea, asthma, tuberculosis, chronic obstructive pulmonary disease, sleep apnea or any other ventilatory / lung disease.
11. Treatment with another investigational drug within 3 months prior to screening or having participated in more than four investigational drug studies within 1 year prior to screening.
12. History of moderate to severe motion sickness.
13. Subjects who are unwilling to remove excessive facial hair preventing sealing of the occlusive face mask.
14. Subjects who, in the opinion of the investigator, will not be able to participate optimally in the study.
15. Any surgical or medical condition which might significantly alter the distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following, and be discussed with the Sponsor prior to enrollment into the trial:

    1. history of pancreatic injury or pancreatitis;
    2. history or presence of liver disease or liver injury;
    3. history of previously elevated ALT/AST values;
    4. history or presence of impaired renal function as indicated by clinically significant elevation in creatinine, BUN/urea, urinary albumin, or clinically significant urinary cellular constituents; or
    5. history of urinary obstruction or difficulty in voiding.
16. Subject who has a history of any infectious disease within 4 weeks prior to drug administration that in the opinion of the investigator, affects the subject's ability to participate in the trial.
17. Subjects who are part of the study staff personnel or family members of the study staff personnel.
18. Subjects who have demonstrated allergic reactions (e.g., food, drug, atopic reactions, or asthmatic episodes) which, in the opinion of the investigator and Sponsor, interfere with their ability to participate in the trial.
19. Subjects who have a history of malignancy and are in remission <5 years.
20. Personal or family history of malignant hyperthermia.
21. Personal or family history of arrhythmias or ECG conductance abnormalities.
22. Subjects with an average daily consumption of a large quantity of coffee, tea, (> 6 cups per day), energy drinks, or equivalent.
23. Subjects with a known history of allergy to lidocaine, xylocaine, or other local anesthetic agents.
24. Subjects with any history of radial-artery (in either arm) disease or injury, or prior known difficulty with placement of arterial line cannula.
25. Subjects with history of known difficult airway access and presence of a "nonreassuring" airway exam (as determined by the investigator), gastroesophageal reflux disease, gastric motility disorders, or delayed gastric emptying.
26. Use of any prescription or over-the-counter medications (such as antacids, vitamins, minerals, dietary/herbal preparations, St. John's Wort, and nutritional supplements) within 14 days prior to Screening; and use of CYP450 inhibitors/inducers within 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Range values of laboratory tests (Safety) | From screening to follow up visit (approx. 8 weeks)
  To determine the safety of single-dose safety of ENA-001 compared to placebo in healthy volunteers after Intravenous (IV) and Intramuscular (IM) injection.
  Primary endpoints include the laboratory range values of safety laboratory tests (hematology, coagulation, clinical chemistry, and urinalysis). Any measurement out of range will be assessed for adverse event.
Range values of special chemistry tests (Safety) | From screening to follow up visit (approx. 8 weeks)
  To determine the safety of single-dose safety of ENA-001 compared to placebo in healthy volunteers after Intravenous (IV) and Intramuscular (IM) injection.
  Primary endpoints include special chemistry assessments (Ca+2 and HCO3- or venous CO2). Any measurement out of range will be assessed for adverse event.
Vital Sign measurements (Safety and tolerability) | From screening to follow up visit (approx. 8 weeks)
  To determine the single-dose safety and tolerability of ENA-001 compared to placebo in healthy volunteers after Intravenous (IV) and Intramuscular (IM) injection.
  Primary endpoints include vital sign measurements (blood pressure and heart rate). Any measurement out of range may indicate an adverse event, meet stopping criteria, and/or indicate intolerability of ENA-001.
  Systolic and diastolic blood pressure (mmHg), pulse rate (HR), body temperature (°C) will be graded according to the FDA guidance Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Measurement of ECG parameters (Safety and tolerability) | From screening to follow up visit (approx. 8 weeks)
  To determine the safety and tolerability of single-dose safety of ENA-001 compared to placebo in healthy volunteers after Intravenous (IV) and Intramuscular (IM) injection.
  Primary endpoints include ECG measurement. Any measurement out of range may indicate an adverse event and/or indicate intolerability of ENA-001.
Complete Physical Exam Findings (Safety and tolerability) | From screening to follow up visit (approx. 8 weeks)
  To determine the safety and tolerability of single-dose safety of ENA-001 compared to placebo in healthy volunteers after Intravenous (IV) and Intramuscular (IM) injection. Primary endpoints include physical examination findings. Complete physical examination will include: head, eyes, ears, nose, throat, neck, heart, chest, lungs, abdomen, extremities, skin, and neurological exam. Any post-baseline findings of the physical examination will be assessed for adverse event.
Incidence of Adverse Events (Safety and tolerability) | From screening to follow up visit (approx. 8 weeks)
  To determine the safety and tolerability of single-dose safety of ENA-001 compared to placebo in healthy volunteers after Intravenous (IV) and Intramuscular (IM) injection. Number of participant with adverse events and grade of AEs will be used to inform on safety and tolerability of ENA-001.

SECONDARY OUTCOMES:
Evaluation of spirometry values (PD) | Each dosing day (Day 1) - Approximately 3 weeks
  To evaluate the single dose pharmacodynamics (PD) of ENA-001 in healthy volunteers after IV and IM dosing. PD will include spirometric measurement for precision in determination of tidal volume (Vt) and respiratory rate (f), which will calculate minute ventilation (MV). These measures are secondary endpoint insomuch as an improvement in ventilation can be seen without a concomitant increase in MV.
Evaluation of capnography values (PD) | Each dosing day (Day 1) - Approximately 3 weeks
  To evaluate the single dose pharmacodynamics (PD) of ENA-001 in healthy volunteers after IV and IM dosing. End-tidal carbon dioxide (ETCO2) reflects the production, transportation, and elimination of CO2. ETCO2 will be monitored by capnography using a suitable patient interface such as a dual O2 delivery and CO2 monitoring cannula. ETCO2 value will be used to determine stopping criteria.
Evaluation of Pulse Oximetry (PD) | Each dosing day (Day 1) - Approximately 3 weeks
  Pulse oximetry: hemoglobin saturation (SpO2) and pulse rate (PR) will determine arterial hemoglobin saturation level in a tissue bed that is reflective of arterial saturation. Continuous decrease in SpO2 and participant will not increase to next dose level.
Evaluation of ABG measurements (PD) | Each dosing day (Day 1) - Approximately 3 weeks
  To evaluate the single dose pharmacodynamics (PD) of ENA-001 in healthy volunteers after IV and IM dosing. Arterial Blood Gases (ABG) values will be used to assess the effectiveness of ventilation. ABG values are precise indicators for interpreting effectiveness of ventilation (pH and PaCO2). ABGs provide ventilation-related data which are independent of minute ventilation (MV). Persistent hyperventilation and associated hypocarbia not relieved by rebreathing exhaled CO2 will be considered a Serious Adverse Event (SAE) and a study stopping criteria.
Evaluation of Cmax (Maximum observed plasma concentration) value (PK) | Each dosing day (Day 1) - Approximately 3 weeks
  Evaluation of single dose pharmacokinetics (PK) of ENA-001 in healthy volunteers after IV and IM dosing. PK parameters of Cmax value greater than specified ng/mL will inform on safety and the subject will meet discontinuation criteria. Data will be assessed by a Safety Review Committee and approval to proceed will be issued prior to subsequent dosing.
Evaluation of AUCinf (Area under the concentration-time curve from time 0 to the time of the last measurable sample) value (PK) | Each dosing day (Day 1) - Approximately 3 weeks
  Evaluation of single dose pharmacokinetics (PK) of ENA-001 in healthy volunteers after IV and IM dosing. PK parameters of AUCinf value greater than specified ng·h/mL will inform on safety and the subject will meet discontinuation criteria. Data will be assessed by a Safety Review Committee and approval to proceed will be issued prior to subsequent dosing.
Evaluation of Tmax (Time to maximum observed plasma concentration) value (PK) | Each dosing day (Day 1) - Approximately 3 weeks
  Evaluation of single dose pharmacokinetics (PK) of ENA-001 in healthy volunteers after IV and IM dosing. PK parameters of Tmax. Data will be assessed by a Safety Review Committee and approval to proceed will be issued prior to subsequent dosing.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dr. Vince Clinical Research, Overland Park, Kansas
  - Clinilabs, Eatontown, New Jersey

IPD SHARING:
Plan to Share IPD: No